CLINICAL TRIAL: NCT04409691
Title: A Clinical Study on the Treatment of Kaposiform Hemangioendothelioma (KHE) With Kasabach-Merritt Phenomenon (KMP) by Hormone Shock and Sirolimus Maintenance
Brief Title: SCMC Trial on KHE With KMP (V.2020)
Acronym: SCMC-KK2020
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCMC2020
Record Dates: First submitted 2020-05-27; First posted 2020-06-01 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Kaposiform Hemangioendothelioma (KHE) With Kasabach-Merritt Phenomenon (KMP)
MeSH Terms: conditions — Kaposiform Hemangioendothelioma | interventions — Sirolimus; Prednisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- prednison group (Active Comparator)
  Interventions: Drug: prednison
- prednison+sirolimus group (Experimental)
  Interventions: Drug: prednison and Sirolimus

INTERVENTIONS:
Drug: prednison and Sirolimus — If the intravenous prednisolone 4 mg / kg / d (one time in the morning and one time in the evening, 2mg / kg body weight each time) is effective, it will be gradually reduced to 2mg / kg / D (one time in the morning and one time in the evening, 1mg / kg body weight each time), gradually converted to oral prednisone of equal dose, and the hormone will be removed within 4-6 weeks. At the same time, the dosage of sirolimus oral liquid is 0.8 mg / m2 twice a day, with an interval of 12 hours, maintaining the blood concentration of 8-15 ng / ml. if there is no intolerable side effect, the treatment will last for 6 months
  Arms: prednison+sirolimus group
Drug: prednison — Prednison is taken at a dose of 4mg/kg/d. If the hormone treatment is effective, it will be gradually reduced to 2mg / kg / d (one time in the morning and one time in the evening, 1 mg / kg body weight each time), and repeated after 2 months of continuous treatment and 1 month of drug withdrawal.
  Arms: prednison group

SUMMARY:
a phase I trial focusing on safety and efficacy of prednison shock plus sirolimus maintenance in treating Kaposiform hemangioendothelioma (KHE) with Kasabach-Merritt phenomenon (KMP)

ELIGIBILITY:
Inclusion Criteria:

* Kaposiform Hemangioendotheliomas with Kasabach-Merritt Phenomenon
* 0 - 12 years of age at the time of study entry
* Male or female
* Consent of parents (or the person having parental authority in families)
* Signed and dated written informed consent

Exclusion Criteria:

* with hematological diseases
* with other solid tumors
* with hypertension, diabetes, adrenal insufficiency, neurological diseases, liver and kidney
* dysfunction, and cardiopulmonary insufficiency
* with tuberculosis,cytomegalovirus and Epstein-Barr virus infection before the treatment

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
response to treatment | 6 months after taking the drug
  Complete Response：
  platelets counts is greater than 100×10^9/L. significant volume reduction is greater than 80%. Fibrinogen levels at 2-4g/L. The surface skin of the tumor is lighter or the tumor is softer significantly.
  Partial Response:
  platelets counts is greater than 40×10^9/L. significant volume reduction is greater than 50%. Fibrinogen levels at less than 50% reduction from baseline. The surface skin of the tumor and palpation of the tumor have no change or less change.
  No Response:
  platelets counts is less than 40×10^9/L. significant volume reduction is less than 50% or the tumor is bigger. Fibrinogen levels at grater then 50% reduction from baseline. The surface skin of the tumor is darker or the tumor is harder.

SECONDARY OUTCOMES:
side effect rate | 6 months after taking the drug
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 Monitoring patient's clinical biochemical indicators and symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Children's Medical Center Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China